CLINICAL TRIAL: NCT00856635
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of the Effects of Glatiramer Acetate (GA) on the Retinal Nerve Fiber Layer (RNFL) and Visual Function in Patients With a First Episode of Acute Optic Neuritis (AON)
Brief Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of the Effects of Glatiramer Acetate (GA) on the Retinal Nerve Fiber Layer (RNFL) and Visual Function in Patients With a First Episode of Acute Optic Neuritis (AON). (Octagon)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM030
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Glatiramer acetate (Experimental): Participants received glatiramer acetate 20 mg subcutaneous injection once a day for up to 6 months.
  Interventions: Drug: Glatiramer Acetate
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once a day for up to 6 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Glatiramer Acetate — 20 mg injected daily subcutaneously
  Other Names: Copaxone
  Arms: Glatiramer acetate
Drug: placebo — injected daily subcutaneously
  Arms: Placebo

SUMMARY:
The main objective of the study is to determine whether glatiramer acetate 20 mg once daily reduces the amount of axonal loss in the optic nerve after a first event of acute optic neuritis compared to placebo patients and to generate data supporting the potential neuroprotective effect of glatiramer acetate in a human in vivo model of axonal loss.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45 years
* Isolated, unilateral, first acute optic neuritis (AON) event consistent with inflammatory demyelinization, not explained by other etiologies. Onset of AON is defined by the presentation of visual disturbances.
* Able to provide written informed consent prior to enrollment
* Willing and able to comply with the protocol requirements for the duration of the study
* For women of child bearing potential:

  * A negative urine pregnancy test o
  * Willing to practice an acceptable method of birth control •
* Willing to receive a steroidal regimen

Exclusion Criteria:

* A diagnosis of clinically definite multiple sclerosis (MS) (Clinically Definite Multiple Sclerosis)
* Current use of any approved disease modifying agents for treatment of MS
* Prior clinical episode of optic neuritis in either eye
* Bilateral AON
* Inability to undergo study evaluations in both eyes
* Known ocular or neurological conditions or abnormalities other than refractive error that impair visual function
* Retrogeniculate visual loss
* Refractive error of greater than +6 or -6 diopters
* Neuromyelitis Optica (Devic's disease)
* Systemic diseases that cause inflammatory optic neuropathy, including but not limited to Sarcoidosis, Systemic lupus erythematosus (SLE), Wegener's Granulomatosis, Syphilis, human immunodeficiency virus (HIV)
* Known ocular conditions that preclude dilation
* Any condition that may interfere with performance of Optical Coherence Tomography (OCT): corneal, lens or fundoscopic abnormality, a co-morbid ocular condition not related to optic neuritis as detected on the OCT reading
* Any condition that precludes administration of Glatiramer Acetate, such as a known history of sensitivity to mannitol
* Diabetes Mellitus Types I or II
* Gastric bypass surgery
* Current use of chemotherapy or radiotherapy
* Treatments that may cause visual loss such as plaquenil, anti-tubercular agents, interferon (IFN)-alpha therapy, monoclonal antibodies Cardiac medications that may affect visual evaluations such as digitalis, amiodarone, quinine
* Ongoing treatment with steroids (for longer than 10 days) within the last 3 months
* Significant or unstable medical, systemic, psychiatric or logistical condition that affects the patient's ability to give informed consent or to complete the study procedures
* Use of an investigational drug within 30 days prior to randomization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Kupersmith, MD, Principal Investigator — Roosevelt Hospital; Peter Calabresi, MD, Principal Investigator — John Hopkins School of Medicine

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glatiramer Acetate | Placebo
Started | 22 | 22
Received Study Drug | 20 | 20
Completed | 12 | 14
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 2 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Serious Adverse Event | 1 | 0
Not completed — Other | 1 | 0
Not completed — Discontinued at Randomization | 2 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all patients who had been randomized to the study and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glatiramer Acetate | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.1) | 34.4 (6.5) | 33.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 2
  Caucasian | 13 | 15 | 28
  Black/African American | 1 | 3 | 4
  Hispanic | 3 | 1 | 4
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Retinal Nerve Fiber Layer Thickness at Baseline and Month 6
Description: Axonal loss in the optic nerve (due to optic neuritis) was assessed by measuring retinal nerve fiber thickness of the affected eye using optical coherence tomography (OCT) at Baseline and Month 6.
Time Frame: Baseline and Month 6
Population: The modified ITT intent-to-treat (mITT) analysis set included all patients who had been randomized to the study, received at least one dose of study drug, had a baseline OCT evaluation, and had at least one non-missing post-baseline OCT evaluation.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Glatiramer Acetate | Placebo
Number analyzed (Participants) | 18 | 18
µm
  Baseline (n=18, 18) | 128.1 (11.9) | 130.5 (8.9)
  Month 6 (n=13, 13) | 89.5 (8.9) | 88.0 (5.5)

2. Secondary Outcome: To Evaluate Changes on Additional OCT Parameters and Other Visual Function and Clinical Parameters.
Time Frame: 6 months
Population: Enrollment did not meet expectations, and target sample sizes were not met. As a results, the secondary outcome was not analyzed. There were no data collected for this outcome; there is no data to analyze.
Arm/Group | Glatiramer Acetate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Glatiramer Acetate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glatiramer Acetate (N=20) | Placebo (N=20)
Drug Hypersensitivity (Immune system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment did not meet expectations, and target sample sizes were not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.